CLINICAL TRIAL: NCT01521637
Title: The Efficacy of Neuromuscular Electrical Stimulation to Attenuate Skeletal Muscle Loss in ICU Patients
Brief Title: The Efficacy of Neuromuscular Electrical Stimulation to Attenuate Muscle Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Dominique Hansen, PhD, Hasselt University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMES2012
Record Dates: First submitted 2012-01-18; First posted 2012-01-31 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Muscle Disuse; Neuromuscular Electrical Stimulation (NMES); Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMES (Experimental): The 'NMES' arm will be treated with NMES.
  Interventions: Procedure: Neuromuscular Electrical Stimulation of m. quadriceps femoris
- No NMES (Sham Comparator): The 'No NMES' arm of the experiment will be sham-treated with NMES. The device will be installed, but not used.
  Interventions: Procedure: Sham-treatment: no NMES

INTERVENTIONS:
Procedure: Neuromuscular Electrical Stimulation of m. quadriceps femoris — Neuromuscular Electrical Stimulation of m. quadriceps femoris by using a commercially available muscle stimulator
  Other Names: Electrical stimulation
  Arms: NMES
Procedure: Sham-treatment: no NMES — Sham comparator
  Other Names: No electrical stimulation; the leg will be sham-treated
  Arms: No NMES

SUMMARY:
Subjects who are hospitalized in the ICU will be included after 24 hours of intubation during their ICU stay. Twice-daily Neuromuscular Electrical Stimulation (NMES) will be performed on one leg for 2x40 min per day to assess muscle fiber size. The investigators hypothesize an attenuated loss in muscle fiber size.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 80 years
* Expected sedated time of >24h

Exclusion Criteria:

* Spinal Cord Injury
* Arterial operaties on the legs
* Local wounds that prohibit NMES
* Chronic use of corticosteroids
* Intake of certain antithrombotic drugs
* Presence of implantable cardioverter defibrillator and/or pacemaker

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in muscle fiber cross sectional area (CSA) | 3 hours before and 12 hours after 10 days of twice-daily NMES
  Muscle fiber cross sectional area (in um2) for type I and II fibers will be analyzed by using immunohistochemistry; the change of muscle fiber CSA over time will be measured

SECONDARY OUTCOMES:
Change in upper leg circumference | 3 hours before and 12 hours after 10 days of twice-daily NMES
  Upper leg circumgerence will be measured; the change of upper leg circumference over time will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Belgium